CLINICAL TRIAL: NCT04018339
Title: Phase I Study of RTA 402 in Obese Adults
Brief Title: A Study of RTA 402 in Obese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RTA 402-010
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Obese Adult Male
Keywords: Bardoxolone Methyl; Obese adult; body weight; body composition
MeSH Terms: conditions — Body Weight | interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTA 402 5mg or 10mg oral administration (Experimental)
  Interventions: Drug: Bardoxolone methyl
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bardoxolone methyl — Bardoxolone methyl 5 mg capsules
  Other Names: RTA 402
  Arms: RTA 402 5mg or 10mg oral administration
Drug: Placebo — Capsules containing an inert placebo
  Arms: Placebo

SUMMARY:
To investigate changes in body weight and body composition in obese adults after repeated oral administration of RTA 402 once daily for 16 weeks, using placebo as a control.

ELIGIBILITY:
Inclusion Criteria:

* Written voluntary informed consent to participate in the study
* Male aged ≥ 20 and < 50 years at the time of consent
* BMI ≥ 25.0 kg/m2 measured at screening
* Waist circumference (umbilical position) ≥ 85 cm measured at screening.
* MRI-measured visceral fat area ≥ 100 cm2 measured at screening

Exclusion Criteria:

* Subjects who have undergone weight control procedures (weight loss medicine, surgical therapy, exercise therapy, bariatric diet, etc.) at a medical institution within 3 months before the screening
* Subjects with conditions requiring treatment other than obesity
* History of cardiac failure (e.g., a prior diagnosis of congestive cardiac failure defined as NYHA class III or IV or a history of hospitalization for cardiac failure)

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 22 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in weight measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months
Changes from baseline in fat mass measured by Dual Energy X-ray Absorption | Through study completion, approximately 6 months
Changes from baseline in lean body mass measured by Dual Energy X-ray Absorption | Through study completion, approximately 6 months
Changes from baseline in skeletal muscle mass index measured by Dual Energy X-ray Absorption | Through study completion, approximately 6 months
Changes from baseline in waist | Through study completion, approximately 6 months
Changes from baseline in grip | Through study completion, approximately 6 months
Changes from baseline in visceral adipose tissue measured by Magnetic Resonance Imaging | Through study completion, approximately 6 months
Changes from baseline in abdominal subcutaneous adipose tissue measured by Magnetic Resonance Imaging | Through study completion, approximately 6 months
Changes from baseline in muscle mass measured by Magnetic Resonance Imaging | Through study completion, approximately 6 months
Changes from baseline in body fat mass measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months
Changes from baseline in segmental muscle mass measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months
Changes from baseline in total body water measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months
Changes from baseline in extracellular water measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months
Changes from baseline in basal metabolic rate measured by Bioelectrical Impedance Analysis | Through study completion, approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bio-Pharmatech Kurume Clinical Pharmacology Clinic, Kurume, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Undecided